CLINICAL TRIAL: NCT07346937
Title: Evaluating the Impact of In-Situ Simulation on Interprofessional Healthcare Team Training: A Randomized Trial
Brief Title: Evaluating the Impact of In-Situ Simulation on Interprofessional Healthcare Team Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Faculty of Medicine of the University of Porto (Unknown); Centro de Simulação da Faculdade de Medicina da Universidade do Porto (Unknown); Hospital Pedro Hispano, ULS Matosinhos (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: In-Situ Simulation
Record Dates: First submitted 2025-12-10; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: in Situ Simulation; Simulation in Training Center
Keywords: In Situ Simulation; Simulation Center; Interprofessional Team Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In Situ Simulation (Experimental): Half of the teams will carry out the scenario in an in-situ context, at the ULS Matosinhos - Pedro Hispano Hospital (ULSM-HPH).
  Interventions: Other: In Situ Simulation
- Simulation Center (Active Comparator): Half of the teams will carry out the scenario in a Simulation Center context, at the Faculty of Medicine, University of Porto (SIMFMUP).
  Interventions: Other: Simulation Center

INTERVENTIONS:
Other: In Situ Simulation — Simulation scenario carried out in situ. The training team will consist of 3 facilitators (who will always be the same throughout the study), with each scenario having only 2 facilitators and the principal investigator.
  Each group will be subjected to the same simulation scenario, the process of which is approximately 60 minutes, divided into: Briefing - 10 min; Scenario Development - 15 minutes; Debriefing - 30/35 min.
  Arms: In Situ Simulation
Other: Simulation Center — Simulation scenario carried out in the Simulation Center. The training team will consist of 3 facilitators (who will always be the same throughout the study), with each scenario having only 2 facilitators and the principal investigator.
  Each group will be subjected to the same simulation scenario, the process of which is approximately 60 minutes, divided into: Briefing - 10 min; Scenario Development - 15 minutes; Debriefing - 30/35 min.
  Arms: Simulation Center

SUMMARY:
Clinical simulation has established itself as an essential methodology in healthcare training, enabling the development of technical and non-technical skills in controlled and safe environments. This study proposes a randomized trial that compares the impact of two learning contexts-a simulation center and the in situ simulation (ISS) environment in the operating room-on the training of interprofessional teams. The aim is to evaluate the effectiveness and efficiency of each context in the acquisition and performance of technical and non-technical skills, as well as participants' perceptions of realism, teamwork, and patient safety. The randomized experimental design reinforces the methodological rigor and internal validity of the results, allowing the identification of important differences between the two approaches. The scarcity of studies on interprofessional simulation in a real clinical context underscores the relevance of this research, which may provide scientific evidence to guide training policies and promote safer, more collaborative practices. It is expected that the results will contribute to improving interprofessional training programs and supporting the systematic integration of ISS in the healthcare field, especially in high-complexity environments.

DETAILED DESCRIPTION:
The increasing complexity of healthcare and the need for a coordinated response among different professionals make interprofessional teamwork an essential element for patient safety and quality of care. In this context, clinical simulation has established itself as a fundamental teaching and learning methodology, allowing the training of technical and non-technical skills in controlled and safe environments. Among the different simulation modalities, in situ simulation (ISS) has gained prominence because it occurs in the clinical context itself, involving real teams and resources of the hospital environment. This approach favors the identification of latent threats to safety and the analysis of workflows and communication in high-pressure scenarios. In addition, ISS has demonstrated a positive impact on safety culture and the performance of multidisciplinary teams. Several studies support that simulation based on interprofessional teams promotes mutual understanding of roles, respect between disciplines, and effective coordination during critical situations. The integration of professionals from different areas in realistic scenarios enhances collaborative learning and strengthens communication, leadership, and decision-making skills, central aspects of Non-Technical Skills (NTS). Despite the available evidence, there is still a gap in the literature regarding the direct comparison between simulation in a training center and ISS in the hospital setting, particularly in the surgical center, an environment characterized by professional interdependence and high technical complexity. Thus, this study proposes a randomized trial comparing the impact of ISS and simulation in a training center on the formation of interprofessional teams. The aim is to systematically evaluate the effect of each context on the acquisition and performance of technical and non-technical skills, as well as on professionals' perception of realism, training effectiveness, and patient safety. This study, therefore, aims to contribute to the development of more effective training strategies based on scientific evidence.

ELIGIBILITY:
Inclusion Criteria:

* Professionals working in the surgical center of ULSM-HPH with at least 6 months of experience in the role.
* Availability to participate in the simulation group assigned to them.

Exclusion Criteria:

* Professionals who do not work in the surgical center.
* Participants who cannot complete all phases of the study due to scheduling or health restrictions.
* Pregnant professionals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Simulation Effectiveness (SET-M) | Immediately after the simulation session (Day 1)
  Measured with Simulation Effectiveness Tool - Modified (SET-M). SET-M is a 19-item tool with a three-point Likert scale that measures effectiveness by capturing student feedback on three domains.
  The higher the score, the more effective the simulation training.
Simulation Effectiveness (ICCAS) | Immediately after the simulation session (Day 1)
  Measured with the Interprofessional Collaborative Competencies Attainment Survey (ICCAS).
  ICCAS is a 20-item self-report tool with a seven-point Likert scale that evaluates the participants' competencies in six dimensions before and after the simulation. Participants complete the tool after simulation training, but rate their abilities twice: once as they recall them before training, and after that training is done.
  The higher the score, the more effective the simulation training.
Simulation Design Evaluation | Immediately after the simulation session (Day 1)
  Evaluated using Simulation Design Scale (SDS) - Student version. SDS is a 20-item tool with a five-point Likert scale designed to evaluate five design features of instructor-developed simulations.
  The instrument has two parts: the presence of specific features in the simulation and the importance of those features to the learner.
  The higher the score, the higher the evaluation of the design feature.
Simulation Debriefing Assessment | Immediately after the simulation session (Day 1)
  Measured with the Debriefing Assessment for Simulation in Healthcare (DASH) Short version for students and for instructors.
  DASH for students has students evaluating the instructors in 6 elements with a seven-point Likert scale, while DASH for instructors is a self-assessment tool with the same structure.
  The higher the score, the higher the debriefing skill.

CONTACTS AND LOCATIONS:
Overall Officials: Maria do Céu F Campos, Principal Investigator — Universidade do Porto
Locations (2):
- Portugal (2):
  - ULS Matosinhos - Hospital Pedro Hispano, Matosinhos Municipality
  - Faculty of Medicine, University of Porto, Porto

IPD SHARING:
Plan to Share IPD: Undecided